CLINICAL TRIAL: NCT04178564
Title: Major Memory 2: A Long-term Group Cognitive Stimulation Program for Patients With Neurocognitive Disorders Attending Social Responses in Oliveira do Bairro Municipality
Brief Title: Major Memory 2: A Long-term Group Cognitive Stimulation Program
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 pandemic
Sponsor: Rsocialform - Geriatria, Lda (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14112019
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Neurocognitive Disorders; Dementia; Cognitive Impairment; Cognitive Decline
Keywords: Neurocognitive Disorders; Dementia; Cognitive Impairment; Cognitive Decline; Elderly; Cognitive Stimulation; Group Intervention; Cognition; Depression
MeSH Terms: conditions — Neurocognitive Disorders; Dementia; Cognitive Dysfunction; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Intervention group will receive 47 sessions of group CS and participate in 3 evaluation sessions. The CS program will last 1 year and each group CS session will last approximately 60 minutes.
  Interventions: Behavioral: Cognitive Stimulation

INTERVENTIONS:
Behavioral: Cognitive Stimulation — The intervention includes 50 sessions, over the course of one year, being that 3 of those sessions will be the pretest, intratest and posttest evaluations. The intervention sessions will last approximately 60 minutes and they will be developed according to the following structure:
  Welcoming to the group (5 minutes) Reality orientation therapy (10 minutes) Main activity (35 minutes) Session evaluation (10 minutes) CS sessions will be conducted in groups. The intervention sessions will include several activities based on different non-pharmacological therapies, whose effectiveness in elderly with neurocognitive disorders has been scientifically proven. Non-pharmacological therapies used encompass therapies such as musictherapy, reminiscence therapy, validation therapy, Montessori method in geriatrics, ADL training, art therapy and the computer software Rehacom.

SUMMARY:
This study aims to evaluate the effect of a long-term group cognitive stimulation (CS) program on the cognitive function of institutionalized elderly people with neurocognitive disorders. The study also aims to assess the program's feasibility in institutions located in the Portuguese town of Oliveira do Bairro.

The investigators propose the realization of a quasi-experimental longitudinal study with a one-group pretest-posttest design. The subjects will participate in CS sessions as part of a group, once a week, for one year, while maintaining their usual care in the institution. The program will have 47 sessions, once per week, with 1 hour each. In each participating institution, one group will be formed. In groups composed by participants with mild neurocognitive disorder, the maximum number will be 10 participants per group, in groups composed by participants with major neurocognitive disorder, the maximum number will be 6 participants per group. In each institution, patients who meet the inclusion and exclusion criteria will be selected to become part of a cognitive stimulation group program.

DETAILED DESCRIPTION:
At this moment, the world is experiencing an unprecedented population aging at a global scale. In 2050, the number of people over 65 years old will more than double from 617 million to 1,6 billion and the percentage of people over 65 years old will grow from 9% to 16%. Portugal is one of the fastest aging countries in the world, 22% of its population is over 65 years of age.

With the increase of the elderly population, new challenges arise such as the increased prevalence of neurocognitive disorders. According with estimates from OCDE, Portugal is the fourth country with the highest number of dementia diagnosis. This brings many social, health and economic costs to our country.

There is evidence that in the earlier stages of neurocognitive disorders, people can learn and improve their cognitive function through interventions, such as cognitive stimulation (CS). There are three types of cognitive intervention to improve cognitive performance: CS, cognitive rehabilitation and cognitive training. Cognitive rehabilitation is an individualized approach to improve cognitive impairment and enhance everyday functioning. Cognitive training is designed for the patient to perform a set of tasks to improve or maintain cognitive function through guided practice.

CS is an intervention where cognitive domains are not used in isolation but in an integrated manner. CS can be structured in an individual or group format. Individual CS therapy includes activities designed to stimulate cognition, conducted only with the therapist and the patient.

On the other hand, group CS is the "engagement in a range of group activities and discussions aimed at general enhancement of cognitive and social functioning".

In a study that applied individual CS therapy in institutionalized Portuguese patients with mild neurocognitive disorder, over the course of one year, it was found a significant improvement in the intervention group on cognitive performance and a significant reduction of depressive symptoms, with medium to large effect sizes, showing that CS therapy is effective in the individual format.

However, CS is also effective when conducted in groups. The results of a group CS therapy program conducted in a multicenter, single blind, randomized controlled trial, showed significant improvements on cognitive performance in the intervention group, specifically in the scores of Mini Mental State Examination and the cognitive subscale of the Alzheimer's Disease Assessment Scale.

Following this evidence, the National Institute for Health and Clinical Excellence has recommended structured Group CS as a non-pharmacological therapy for people with mild to moderate neurocognitive disorder.

In a systematic review about CS, studies showed strong evidence that CS has a positive impact on cognitive performance, depression, activities of daily living and behavior for people with neurocognitive disorders.

In a multicenter study conducted with a one-group design and 14 group CS sessions over the course of 7 weeks, in patients with mild to moderate dementia, results showed an improvement on cognitive domains, such as memory, language comprehension and orientation, but did not show significant changes on attention/working memory, executive function or praxis.

In another study, which involved conducting a 10 session cognitive stimulation program, each session lasting 2 hours, 3 times per week, with elderly living in social protection centers, it was also found a statistically significant improvement in the participants' cognitive functioning after the intervention.

Another study involved a multicenter investigation where a group CS program was applied to people with diagnosis of mild to moderate dementia. The program was based on the Making a Difference program of Spector et al. which has 14 bi-weekly sessions, over the course of 7 weeks. Results showed a significant improvement on cognitive functions and also in depressive symptomatology.

In a study carried out in Portugal, a group CS program for people with mild cognitive impairment, composed by 1 weekly session, lasting 90 minutes, for 8 weeks, obtained positive results. It concluded that short term memory, orientation, language and visuospatial orientation improved significantly in the intervention group in comparison with the control group.

Other portuguese authors also applied a group CS program, which was based on the Making a Difference Program, with 14 twice a week sessions, each lasting 45-60 minutes. This study found a significant improvement on cognitive functions in the participants of the intervention group.

Considering the previous information, this research proposition's goal is to evaluate the effect of group CS on cognitive performance and depressive symptomatology in institutionalized people with mild to major neurocognitive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of neurocognitive disorder according to the Diagnostic and Statistical Manual of Mental Disorder.
* Having a score between 2 and 5 according to the Global Deterioration Scale (obtained from the participant's score on Mini-Mental State Examination).
* Age over 60 years old.
* Attending one of the institutions participating in the study.

Exclusion Criteria:

* To have received psychological or psychiatric care in the last two months.
* Not being able to communicate and understand.
* To suffer from an acute or severe illness that makes their participation in the sessions impossible.
* Sensory and physical limitation that prevent their participation in the sessions.
* Limited attention span that prevents attending a one-hour group session.
* Presence of severe neuropsychiatric symptoms that prevent their participation in the sessions or uncontrolled delirium.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive functioning evaluated through Mini-Mental State Examination | Time Frame: Pre, intra (6 months) and post intervention (12 months)
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and post-intervention assessments. Mini-Mental State Examination is a brief screening test for cognitive function. Assesses 6 cognitive functions: orientation, registration, attention and calculation, recall, language and visuoconstructive ability. Global score ranges from 0-30 points, higher scores indicate better cognitive function.
Cognitive functioning evaluated through Frontal Assessment Battery | Time Frame: Pre, intra (6 months) and post intervention (12 months)
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and post-intervention assessments. Frontal Assessment Battery is a screening test for executive functioning. Assesses conceptualization, lexical fluency, programming or motor series, sensitivity to interference, inhibitory control and environmental autonomy. Each subtest is scored from 0-3 points and global score ranges from 0-18 points. A higher score indicates a better executive function.

SECONDARY OUTCOMES:
Mood evaluated through Geriatric Depression Scale -15 | Time Frame: Pre, intra (6 months) and post intervention (12 months)
  Significant statistic improvement in the participant's test scores between pre-intervention, intra-intervention and post-intervention assessments. Geriatric Depression Scale -15 is a screening test for depressive symptoms in elderly adults. Assesses depression in the elderly by distinguishing between depressive and dementia symptoms. This instrument does not include somatic conditions common to the elderly, such as apetite, sleep or sexual disturbances, or lower energy level. The overall score ranges from 0 to 15. The higher the score, the greater the severity of the depressive symptoms.

OTHER OUTCOMES:
Sociodemographic data collected through a sociodemographic questionnaire | Time Frame: Pre-intervention
  Sociodemographic data will be collected using a sociodemographic questionnaire, designed specifically for this study, regarding information about age, gender, literacy, health conditions, among others.
Adherence to the intervention and dropouts evaluated through a session form | Time Frame: Pre, intra (6 months) and post intervention (12 months)
  Adherence to the intervention and dropouts will be assessed using a session form, designed specifically for this study, completed by the technician after each session, regarding the attendance and mood/behavior of the participants throughout the intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Susana I Justo Henriques, PhD, Principal Investigator — Replicar Socialform and University of de Santiago de Compostela; Patricia Otero Otero, PhD, Principal Investigator — Universidade da Coruña; Vanessa Blanco Seoane, PhD, Principal Investigator — University of de Santiago de Compostela; Fernando L Vázquez González, PhD, Principal Investigator — University of de Santiago de Compostela
Locations (8):
- Portugal (8):
  - Rsocialform - Geriatria, Lda., Mealhada, Aveiro District
  - Associação de Solidariedade Social do Silveiro, Oliveira do Bairro
  - Associação dos Amigos de Perrães, Oliveira do Bairro
  - Centro Ambiente para Todos, Oliveira do Bairro
  - Centro Social de Oiã, Oliveira do Bairro
  - Centro Social Paroquial de S.Pedro da Palhaça, Oliveira do Bairro
  - Santa Casa da Misericórdia de Oliveira do Bairro, Oliveira do Bairro
  - Sóbustos, Oliveira do Bairro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apostolo JL, Cardoso DF, Rosa AI, Paul C. The effect of cognitive stimulation on nursing home elders: a randomized controlled trial. J Nurs Scholarsh. 2014 May;46(3):157-66. doi: 10.1111/jnu.12072. Epub 2014 Mar 5. PMID 24597922
- [Background] Apóstolo JL, Loureiro LMJ, Carvalho IA, Alves I, Batista DF, Sfetcu R. Contribution to the adaptation of the Geriatric Depression Scale -15 into Portuguese. Revista de Enfermagem Referencia 3: 65-73, 2014. doi:10.12707/RIV14033
- [Background] Apóstolo JLA, Bobrowicz-Campos EM, dos Reis IAC, Henriques SJ, Correia CAV. Exploring the screening capacity of the European Portuguese version of the 15-item Geriatric Depression Scale. Revista de Psicopatología y Psicología Clínica 23: 99-107, 2018. doi: 10.5944/rppc.vol.23.num.2.2018.21050
- [Background] Clare L, Wilson BA, Carter G, Breen K, Gosses A, Hodges JR. Intervening with everyday memory problems in dementia of Alzheimer type: an errorless learning approach. J Clin Exp Neuropsychol. 2000 Feb;22(1):132-46. doi: 10.1076/1380-3395(200002)22:1;1-8;FT132. PMID 10649552
- [Background] Clare L, Woods RT. Cognitive training and cognitive rehabilitation for people with early-stage Alzheimer's disease: a review. Neuropsychological Rehabilitation 14: 385-401, 2004
- [Background] Costa ARD, Sequeira C. Efetividade de um Programa de Estimulação Cognitiva em Idosos com Défice Cognitivo Ligeiro. Revista Portuguesa de Enfermagem de Saúde Mental 9: 14-20, 2013
- [Background] Davis RN, Massman PJ, Doody RS. Cognitive intervention in Alzheimer disease: a randomized placebo-controlled study. Alzheimer Dis Assoc Disord. 2001 Jan-Mar;15(1):1-9. doi: 10.1097/00002093-200101000-00001. PMID 11236819
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Filipin F, Feldman M, Taragano FE, Martelli M, Sánchez V, García V, Tufro G, Heisecke S, Serrano C, Dillon, C. The Efficacy of Cognitive Stimulation on Depression and Cognition in Elderly Patients with Cognitive Impairment: A Retrospective Cohort Study. AIMS Medical Science 3 (1): 1-14, 2015
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Freitas S, Simoes MR, Alves L, Santana I. The Relevance of Sociodemographic and Health Variables on MMSE Normative Data. Appl Neuropsychol Adult. 2015;22(4):311-9. doi: 10.1080/23279095.2014.926455. Epub 2014 Dec 22. PMID 25531579
- [Background] Guerreiro M, Silva AP, Botelho MA, Leitão O, Castro-Caldas A, Garcia C. Adaptação à população portuguesa da tradução do Mini Mental State Examination (MMSE). Revista Portuguesa de Neurologia 1 (9): 9-10, 1994
- [Background] Hall L, Orrell M, Stott J, Spector A. Cognitive stimulation therapy (CST): neuropsychological mechanisms of change. Int Psychogeriatr. 2013 Mar;25(3):479-89. doi: 10.1017/S1041610212001822. Epub 2012 Nov 12. PMID 23146408
- [Background] Justo-Henriques SI, Marques-Castro AE, Otero P, Vazquez FL, Torres AJ. [Long-term individual cognitive stimulation program in patients with mild neurocognitive disorder: a pilot study]. Rev Neurol. 2019 Apr 1;68(7):281-289. doi: 10.33588/rn.6807.2018321. Spanish. PMID 30906977
- [Background] Lima CF, Meireles LP, Fonseca R, Castro SL, Garrett C. The Frontal Assessment Battery (FAB) in Parkinson's disease and correlations with formal measures of executive functioning. J Neurol. 2008 Nov;255(11):1756-61. doi: 10.1007/s00415-008-0024-6. Epub 2008 Sep 25. PMID 18821046
- [Background] Lobbia A, Carbone E, Faggian S, Gardini S, Piras F, Spector A, Borella E. The efficacy of cognitive stimulation therapy (CST) for people with mild-to-moderate dementia: A review. European Psychologist, 2018. doi:10.1027/1016-9040/a000342
- [Background] Loewenstein DA, Acevedo A, Czaja SJ, Duara R. Cognitive rehabilitation of mildly impaired Alzheimer disease patients on cholinesterase inhibitors. Am J Geriatr Psychiatry. 2004 Jul-Aug;12(4):395-402. doi: 10.1176/appi.ajgp.12.4.395. PMID 15249277
- [Background] Melguizo Herrera E, Bertel De La Hoz A, Paternina Osorio D, Felfle Fuentes Y, Porto Osorio L. Cognitive Stimulation of Elderly Residents in Social Protection Centers in Cartagena, 2014. Rev Colomb Psiquiatr. 2017 Oct-Dec;46(4):229-236. doi: 10.1016/j.rcp.2016.09.008. Epub 2016 Nov 2. PMID 29122230
- [Background] Morgado J, Rocha CS, Maruta C, Guerreiro M, Martins IP. Novos valores normativos do Mini-Mental Sate Examination. Sinapse 2 (9): 10-16, 2009
- [Background] Sheikh JI, Yesavage JA. Geriatric Depression Scale (GDS): Recent evidence and development of a shorter version. Clinical Gerontologist: The Journal of Aging and Mental Health 5 (1-2): 165-173, 1986
- [Background] Spector A, Thorgrimsen L, Woods B, Royan L, Davies S, Butterworth M, Orrell M. Efficacy of an evidence-based cognitive stimulation therapy programme for people with dementia: randomised controlled trial. Br J Psychiatry. 2003 Sep;183:248-54. doi: 10.1192/bjp.183.3.248. PMID 12948999
- [Background] Wilson B. Towards a comprehensive model of cognitive rehabilitation. Neuropsychol Rehabil 12: 97-110, 2002
- [Background] Woods B, Aguirre E, Spector AE, Orrell M. Cognitive stimulation to improve cognitive functioning in people with dementia. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD005562. doi: 10.1002/14651858.CD005562.pub2. PMID 22336813
- [Background] Reisberg B, Ferris SH, de Leon MJ, Crook T. The Global Deterioration Scale for assessment of primary degenerative dementia. Am J Psychiatry. 1982 Sep;139(9):1136-9. doi: 10.1176/ajp.139.9.1136. PMID 7114305